CLINICAL TRIAL: NCT01442337
Title: A Phase 2/3, Double-Blind, Placebo-Controlled, Two-Part Study (Part 1 Open-Label) to Assess the Safety, Efficacy and Pharmacokinetics of Single Intravenous Doses of ASP8597 (Diannexin) in de Novo Kidney Transplant Recipients
Brief Title: A Study to Evaluate the Effect of ASP8597 in Adult Kidney Transplant Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was terminated by sponsor decision
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 8597-CL-0201
Record Dates: First submitted 2011-09-16; First posted 2011-09-28 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Kidney Transplantation
Keywords: de novo kidney transplant; kidney transplant; ASP8597; diannexin; ischemia-reperfusion injury
MeSH Terms: conditions — Reperfusion Injury | interventions — diannexin, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ASP8597 low dose (Experimental)
  Interventions: Drug: ASP8597
- ASP8597 high dose (Experimental)
  Interventions: Drug: ASP8597
- ASP8597 highest dose (Experimental)
  Interventions: Drug: ASP8597
- Placebo (Placebo Comparator): Placebo comparator used in Part 2 only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP8597 — one time IV dose
  Other Names: diannexin
  Arms: ASP8597 high dose; ASP8597 highest dose; ASP8597 low dose
Drug: Placebo — one time IV dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of a single intravenous dose of ASP8597 in kidney transplant recipients.

DETAILED DESCRIPTION:
This is a two-part study. Part 1 (Phase 2) has completed enrollment. Subjects are currently being followed per protocol. Data from Part 1 will be used to determine the doses used in Part 2 (Phase 3). Part 2 will enroll approximately 573 subjects and is planned to have 2 doses of ASP8597 (low dose and either the high or highest dose) along with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled to receive a kidney transplant from a deceased donor meeting at least one of the following criteria:

  1. Expanded Criteria Donor (ECD)

     * i Donor was > 60 years of age, OR
     * ii. Donor was 50-59 years of age, inclusive, and met at least two of the following criteria:

       1. Donor died of a cerebral bleed
       2. Donor had a history of hypertension
       3. Donor's terminal serum creatinine concentration was > 1.5 mg/dL
  2. Donation after Cardiac Death (DCD) - Donor was pronounced dead prior to procurement of the kidney
  3. Standard Criteria Donor (SCD)

     * i. Donor with terminal serum creatinine < 1.5 mg/dL where kidney is anticipated to have a minimum of 24 hours of cold ischemia prior to transplantation, OR
     * ii. Donor with terminal serum creatinine > 1.5 mg/dL and any cold ischemic time up to exclusion limit
* Female subject is not pregnant and agrees to use an acceptable form of contraception throughout study
* Male subject agrees to use an adequate method of contraception and agrees to no sperm donation throughout the study

Exclusion Criteria:

* Female subject is pregnant or lactating
* Donor kidney is anticipated to have more than 40 hours of cold ischemia time
* Donor is > 66 years of age
* Donor meets both DCD and ECD criteria
* Subject has previously received, or is receiving an organ transplant other than a kidney
* Subject has a positive T or B cell crossmatch by the investigational site's standard method of determination. For recipients where only a flow cytometry crossmatch is performed and is positive in either T or B cell testing, recipients are excluded only if donor specific, anti-HLA antibody is detected by flow cytometry based, specific anti-HLA antibody testing
* Subject has ABO blood type incompatibility with his/her organ donor
* Recipient or donor is known by medical history to be seropositive for human immunodeficiency virus (HIV)
* Subject has a known bleeding diathesis
* Subject has a International Normalized Ratio (INR) > 1.5 times upper limit of normal at Screening
* Subject has a platelet count < 100,000 platelets/µL at Screening
* Subject used anti-platelet agents [e.g., Plavix® (clopidogrel bisulfate), Brilinta® (ticagrelor)] (with the exception of aspirin < 100 mg/day for cardiovascular prophylaxis), anti-coagulants [e.g., Pradaxa® (dabigatran), Xarelto® (rivaroxaban)], anti-thrombotics, and/or blood-thinning agents within the 10 days prior to Screening; and/or subject is expected to require use of any of these agents during the first 15 days of the study period (with the exception of standard of care peri-operative administration of heparin for DVT prophylaxis)
* Subject has an uncontrolled concomitant infection
* Subject has a current malignancy or a history of any malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully
* Subject currently is participating in an investigational drug study, or participated in an investigational drug study within the last 30 days)
* Subject has a history of or is believed to have used an illicit drug(s) and/or abused alcohol within the last 3 months
* Subject has an unstable psychiatric illness
* Subject has previously received ASP8597 or participated in a study involving ASP8597

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) variable for ASP8597: Maximum concentration (Cmax) | 3 days
  Part 1 PK variable
Pharmacokinetic variable for ASP8597: Area under the concentration-time curve from time 0 to last quantifiable concentration (AUClast) | 3 days
  Part 1 PK variable
Pharmacokinetic variable for ASP8597: Area under the concentration-time curve from time 0 to infinity (AUCinf) | 3 days
  Part 1 PK variable
Estimated glomerular filtration rate (eGFR) using abbreviated Modified Diet in Renal Disease (MDRD) formula - Part 2 | 12 months
  Part 2 efficacy variable

SECONDARY OUTCOMES:
Pharmacokinetic variable for ASP8597: Time to attain Cmax (Tmax) | 3 days
  Part 1 PK variable
Pharmacokinetic variable for ASP8597: Clearance (CL) | 3 days
  Part 1 PK variable
Pharmacokinetic variable for ASP8597: Volume of Distribution (Vz) | 3 days
  Part 1 PK variable
Pharmacokinetic variable for ASP8597: Apparent terminal elimination half-life (t1/2) | 3 days
  Part 1 PK variable
Requirement of dialysis within the first 7 days post transplant - Part 1 | 7 days
  Part 1 efficacy variable
eGFR using abbreviated MDRD formula - Part 1 | 12 months
  Part 1 efficacy variable
Requirement of dialysis within the first 7 days post transplant - Part 2 | 7 days
  Part 2 efficacy variable
Patient survival | 12 months
  Part 2 efficacy variable
Graft survival | 12 months
  Part 2 efficacy variable
Biopsy-proven acute rejection (BPAR) | 12 Months
  Part 2 efficacy variable
Clinically treated rejection | 12 months
  Subjects who receive immunosuppressive medications for the treatment of suspected or biopsy-proven acute rejection. Part 2 efficacy variable

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (19):
- United States (19):
  - St. Vincent Medical Center, Los Angeles, California
  - Sharp Memorial, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of California at San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - St. Barnabas Medical Center, Livingston, New Jersey
  - New York Presbyterian Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Pinnacle Health at Harrisburg, Harrisburg, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin